CLINICAL TRIAL: NCT01942369
Title: A Multi-centre, Prospective, Non-interventional Study to Describe the Efficacy of a Continuous up to 24-week Treatment of Diphereline 3.75mg Following Conservative Surgery in Deep Infiltrating Endometriosis (DIE) Patients Over a Period of 24 Months.
Brief Title: A Study to Describe the Efficacy of Diphereline Following Conservative Surgery in Deep Infiltrating Endometriosis (DIE) Patients Over a Period of 24 Months
Acronym: DIE-NIS
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52014-210
Record Dates: First submitted 2013-09-10; First posted 2013-09-16 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Deep Infiltrating Endometriosis (DIE)
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Triptorelin Pamoate; Injections, Intramuscular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deep Infiltrating Endometriosis (DIE)
  Interventions: Drug: Triptorelin Acetate 3.75mg intramuscular injection

INTERVENTIONS:
Drug: Triptorelin Acetate 3.75mg intramuscular injection — Triptorelin Acetate is a Gonadotrophin Releasing Hormone agonist (GnRHa).
  Triptorelin acetate for injection 3.75mg administered as described in the patient information sheet approved in China: one intramuscular injection of the product repeated every 4 weeks.
  Other Names: Diphereline 3.75mg intramuscular injection

SUMMARY:
The purpose of this study is to describe changes in the intensity of specific endometriosis symptoms from baseline pre-surgery to after surgery and subsequent continuous Diphereline (Triptorelin Acetate) treatment for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DIE and having received surgery treatment within one month before inclusion
* Premenopausal women aged >=18 years old.
* Written ICF has been obtained prior to any study-related procedures
* Patient for whom the treating physician already made the decision to treat by Diphereline.
* Patient should be mentally and physically able to express her symptom complaints and answer questions.

Exclusion Criteria:

* Pregnancy or lactation.
* Patients currently on treatment or who have been on therapy with a GnRHa in the last 6 months.
* Premenopausal women who may reach menopause within the 3 years post randomisation.
* Hypersensitivity to Triptorelin or one of the excipients of Triptorelin 3.75mg
* Treatment with another research drug over the last 3 months before the study
* Potentially unreliable patients, and those judged by the investigator to be unsuitable for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital patients who had been diagnosed with DIE, surgically treated and for whom decision has been made to be treated with a GnRHa post-surgery.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2013-09-16; Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Changes in the intensity of specific endometriosis symptoms from baseline pre-surgery | Every 3 months in the first 12 months after surgery and every 6 months in the following 12 months
  The specific endometriosis symptoms include pelvic pain, dysmenorrhoea, pain at time of ovulation, dyspareunia to be assessed with a 10-cm visual analogue scale (VAS).
  Other symptoms (Amenorrhea, menorrhagia, metrorrhagia, Global GI symptoms & urinary discomfort,) will be assessed by oral enquiry to the patients based on numerical scale from 0 to 10 (0 being the best and 10 the worst status).

SECONDARY OUTCOMES:
Recurrence rate of specific endometriosis symptoms | At 12 months and 24 months
  Recurrence rate of specific endometriosis symptoms in the group of patients with mild or null symptoms score following surgery and Diphereline treatment.
Change during the study period in symptom(s) having the highest intensity at baseline | 24 months
  The highest intensity at baseline is defined as the symptom with the highest score on pre-surgery assessment.
Rate of pregnancy in subjects | At 12 months and 24 months
Abdominal pain-free interval | Every 3 months in the first 12 months after surgery and every 6 months in the following 12 months
  Assessed using a visual analogue scale (VAS).
Disease profile of DIE patients treated by Diphereline and by duration of treatment. | 24 months
  The disease profile (size of the lesion, locations etc…) will be detailed in each group of treatment duration by descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (18):
- China (18):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Jishuitan Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Xinqiao Hospital,Third Military Medical University, Chongqing
  - Southwest Hospital,Chongqing,400038, Chongqing
  - Women's Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Anhui Provincial Cancer Hospital,Hefei,China,230031, Hefei
  - Jiangxi Maternal and Child Health Hospital,Nanchang, Nanchang
  - Nanjing Maternity and Child Health Care Hospital, Nanjing
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai
  - The International Peace Maternity & Child Health Hospital of China, Shanghai
  - Shanghai First Maternity and Infant Hospital, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - The Second Hospital of Shanxi Medical University,Taiyuan, Taiyuan
  - Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University (Hubei General Hospital), Wuhan
  - Henan Provincial People's Hospital, Zhengzhou

REFERENCES:
- [Derived] Zhu L, Guan Z, Huang Y, Hua K, Ma L, Zhang J, Yang D, Perrot V, Li H, Zhang X. The efficacy and safety of triptorelin-therapy following conservative surgery for deep infiltrating endometriosis: A multicenter, prospective, non-interventional study in China. Medicine (Baltimore). 2022 Feb 4;101(5):e28766. doi: 10.1097/MD.0000000000028766. PMID 35119037
- [Derived] Sun W, Hua K, Hong L, Zhang J, Hao M, Wang J, Zhang J, Perrot V, Li H, Zhang X. Symptom control after different duration of triptorelin treatment following conservative surgery for deep infiltrating endometriosis: Post-hoc analysis of a multicentre, prospective, real-world study. Medicine (Baltimore). 2021 Jul 30;100(30):e26753. doi: 10.1097/MD.0000000000026753. PMID 34397719